CLINICAL TRIAL: NCT01182038
Title: The Swedish Birth Seat Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsingborgs Hospital (Other)
Collaborators: The Stig & Ragna Gorthon Foundation, Helsingborg (Unknown)
Responsible Party: Li Thies-Lagergren, MMid, Reg. Midwife, Reg. Nurse, Doctoral student, The Karolinska Institute, Stockholm and Helsingborgs Hospital, Sweden.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2009/739
Record Dates: First submitted 2010-08-10; First posted 2010-08-16 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Instrumental Vaginal Births; Oxytocin Augmentation for Labor; Maternal Blood Loss; Perineal Outcomes; Fetal Outcomes
Keywords: birth seat; childbirth; instrumental delivery; upright position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Birth seat group (Experimental): Randomized to birth on a midwife designed birth seat
  Interventions: Device: BirthRite birthing seat
- Non-birth seat group (No Intervention): Randomized to birth in any other position except on the midwife designed birth seat.

INTERVENTIONS:
Device: BirthRite birthing seat — Randomization takes place on admission to the labor ward when the participants are in active labor.Participants in this arm were to sit on the seat for 20 minute periods.After these 20 minutes, the participant should stand and mobilize during two to three contractions, before resuming the birth seat position. If progress of the descent of the fetal head was obvious the participant was not asked to mobilize.
  Other Names: BirthRite® birthing seat
  Arms: Birth seat group

SUMMARY:
The purpose of this study is to determine whether birth on a birthing seat will effect numbers of instrumentally assisted vaginal births, vaginal traumas, blood loss,use of artificial oxytocin for labour augmentation and fetal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous women who understood the Swedish language sufficiently well to receive information and give informed consent
* a normal pregnancy,singleton fetus in cephalic presentation
* spontaneous onset of labor occurring between gestational weeks 37 + 0 and 41 + 6
* Body Mass Index less (BMI) than thirty
* gestational diabetes not requiring medical treatment
* women who were planning a vaginal birth after a caesarean section (VBAC)
* women induced because of spontaneous rupture of membranes with no spontaneous contractions for longer than twenty-four hours

Exclusion Criteria:

* multiparous women
* birth before gestational week 37
* breech presentation
* maternal BMI more than 30
* multiple pregnancy
* infectious disease
* pre-eclampsia or other conditions requiring medical care

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1002 (Actual)
Dates: Start 2007-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Instrumental vaginal births | Recorded within 6 hours postpartum
  Instrumental births include vacuum extraction and forceps delivery.

SECONDARY OUTCOMES:
Administration of oxytocin for augmentation of labor | During labor and birth up to 36 hours postpartum
Postpartum blood loss | Up to 24 hours after birth
  Blood loss postpartum is weighed and measured and maternal hemoglobin levels are registered.
Perineal outcomes | Up to 36 hours after birth
  Perineal outcomes include vaginal and perineal traumas, episiotomies and perineal edema.
Fetal outcomes | Up to 36 hours after birth
  Fetal outcomes include Apgar scores, cord blood pH levels and admissions to the NICU.

CONTACTS AND LOCATIONS:
Overall Officials: Ingegerd Hildingsson, PhD, Study Director — Karolinska Institutet; Linda J Kvist, PhD, Study Chair — Helsingborg Hospital, Sweden
Locations (1):
- Helsingborgs Hospital, Helsingborg, Skåne County, Sweden

REFERENCES:
- [Derived] Thies-Lagergren L, Kvist LJ, Christensson K, Hildingsson I. Striving for scientific stringency: a re-analysis of a randomised controlled trial considering first-time mothers' obstetric outcomes in relation to birth position. BMC Pregnancy Childbirth. 2012 Nov 22;12:135. doi: 10.1186/1471-2393-12-135. PMID 23173988
- [Derived] Thies-Lagergren L, Kvist LJ, Christensson K, Hildingsson I. No reduction in instrumental vaginal births and no increased risk for adverse perineal outcome in nulliparous women giving birth on a birth seat: results of a Swedish randomized controlled trial. BMC Pregnancy Childbirth. 2011 Mar 24;11:22. doi: 10.1186/1471-2393-11-22. PMID 21435238